CLINICAL TRIAL: NCT00951054
Title: A Phase II Study of NK012 in Locally Advanced Non-Resectable and Metastatic Breast Cancer Patients With Triple Negative Phenotype
Brief Title: A Study of NK012 in Patients With Advanced, Metastatic Triple Negative Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nippon Kayaku Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A6012211US
Record Dates: First submitted 2009-05-21; First posted 2009-08-04 (Estimated); Last update posted 2015-02-16 (Estimated); Status verified 2015-02

CONDITIONS: Triple Negative Breast Cancer
Keywords: breast cancer; triple negative; ER-negative; PR-negative; HER2-negative; ER-, PR-, HER2- (Triple Negative) breast cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: NK012 — 30 minute IV infusion once every 28 days. NK012 dose is 28 mg/m^2 (or 18 mg/m^2 depending on UGT1A1 polymorphism, with potential to dose escalate). Dose escalation cannot exceed 28 mg/m^2. Dosing will proceed until progression or unacceptable toxicity develops, or decision by patient or investigator to stop.

SUMMARY:
The purpose of this study is to determine whether NK012 is safe and effective in the treatment of advanced and metastatic triple negative breast cancer.

DETAILED DESCRIPTION:
This is a Phase II, open label, single arm, multicenter study of NK012 in patients with locally advanced non-resectable and metastatic breast cancer with ER-negative, PR negative and HER2-negative phenotype. NK012 will be administered by infusion over 30 minutes once every 28 days (on Day 1 of each cycle). Patients will be screened for UGT1A1 polymorphism prior to enrollment in order to determine their starting dose.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of breast cancer with locally advanced disease for which there is no surgical option, or stage IV disease.
* ER-negative and PR-negative (defined as less than or equal to 10% tumor staining).
* HER2-negative defined as one of the following:

  1. 0 or 1+ IHC;
  2. 2+ or 3+ IHC and FISH negative (ratio < 2.2);
  3. or FISH negative (ratio < 2.2).
* No less than one and no more than two prior chemotherapy regimens for advanced or metastatic disease.
* Prior chemotherapy must have included a taxane either as part of an adjuvant regimen or as part of a metastatic disease regimen.
* Interval from last dose of prior treatment to enrollment in this study must be at least 4 weeks for cytotoxic chemotherapy (exception: 6 weeks for nitrosoureas or mitomycin C), 5 half-lives for non-cytotoxic therapy (to be reviewed by the Medical Monitor to establish start date), and 4 weeks for monoclonal antibodies; patients must have recovered from all acute toxicities.
* Measurable disease by RECIST.
* ECOG performance status of 0-2.
* Females at least 18 years of age.
* Adequate bone marrow function as defined by absolute neutrophil count of greater than or equal to 1,500/ mm^3 and platelets of greater than or equal to 100,000/mm^3.
* AST(SGOT) and ALT(SGPT) levels no greater than 3 x the institutional ULN, and total bilirubin less than or equal to 1.5 x ULN.
* Serum creatinine less than or equal to 1.5 x ULN, or creatinine clearance greater than or equal to 60 mL/min (Cockcroft-Gault formula) for patients with serum creatinine levels > 1.5 x ULN.
* Able to understand and show willingness to sign a written informed consent document.

Exclusion criteria:

* Patient has Gilbert's Syndrome.
* Concurrent use of other investigational agent.
* History of brain metastases or spinal cord compression, unless irradiated a minimum of 4 weeks before study entry and stable without requirement for corticosteroids for > 1 week.
* Prior exposure to topoisomerase 1 inhibitors (i.e., irinotecan, topotecan, camptothecin).
* Concurrent serious infections requiring parenteral therapy.
* Pregnant or of childbearing potential and not using methods to avoid pregnancy. A negative pregnancy test (urine or serum) must be documented at baseline for women of childbearing potential. Patients may not breast-feed infants while on this study.
* Significant cardiac disease including heart failure that meets New York Heart Association (NYHA) class III and IV definitions, history of myocardial infarction within one year of study entry, uncontrolled dysrhythmias or poorly controlled angina.
* History of serious ventricular arrhythmia (VT or VF, greater than or equal to 3 beats in a row), QTc greater than or equal to 450 msec for men and 470 msec for women, or LVEF less than or equal to 40% by MUGA or ECHO.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Estimated)
Dates: Start 2009-02; Primary Completion 2014-12 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Antitumor activity (overall response rate) of NK012 | At baseline and after every 2 cycles; PR or CR must be confirmed no less than 4 weeks after the first response was recorded

SECONDARY OUTCOMES:
Duration of response | Monthly for 6 months after patient goes off study, then every 3 months thereafter
Rate and duration of disease control | Monthly for 6 months after patient goes off study, then every 3 months thereafter
Time to disease progression | Monthly for 6 months after patient goes off study, then every 3 months thereafter
Toxicity profile of NK012 | Duration of study, and up to 30 days after discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Denise A Yardley, MD, Principal Investigator — SCRI Development Innovations, LLC
Locations (1):
- Sarah Cannon Research Institute, Nashville, Tennessee, United States